CLINICAL TRIAL: NCT00215085
Title: Cardiac Tumors in Children
Status: Terminated | Type: Observational
Why Stopped: insufficient data
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-091
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Heart Disease
Keywords: pediatric health; cardiac; cardiac tumor; children
MeSH Terms: conditions — Heart Defects, Congenital; Heart Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to define the natural history of untreated cardiac tumors, study the pathology of primary cardiac tumors, review the surgical treatment and results of primary cardiac tumors and to determine the prognosis for these tumors.

DETAILED DESCRIPTION:
Primary cardiac tumors in children are extremely rare. Benign tumors are typically myxomas, lipomas, and rhabdomyomas, while malignant tumors are typically angiosarcomas and rhabdomyosarcomas. Due to the rarity of these tumors, it is difficult to gather meaningful information regarding their natural history, pathology and treatment.

The primary aims are to define the natural history of untreated cardiac tumors, study the pathology of primary cardiac tumors, review the surgical treatment and results of primary cardiac tumors and to determine the prognosis for these tumors. The secondary aims are to discover patterns and consistencies among primary cardiac tumors and to define the best treatment options for these patients. The study will be conducted through a retrospective chart review of about 70 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the congenital surgery database
* Children who have been treated for a primary cardiac tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the congenital surgery database
  * Children who have been treated for a primary cardiac tumor
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2005-05; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States